CLINICAL TRIAL: NCT00424281
Title: Pharmacokinetics of Fondaparinux (Arixtra) to Critically Ill Patients on Vasopressor Therapy
Brief Title: Effectiveness of Blood Clot Medication With Concomitant Blood Pressure Medication
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Collaborators: GlaxoSmithKline (Industry)
Other Study IDs: WSU protocol ID= 066706MP4F
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Last update posted 2007-01-19 (Estimated); Status verified 2007-01

CONDITIONS: ICU Patients 18 Years or Older.
Keywords: Arixtra, fondaparinux, vasopressor, venous thrombolism
MeSH Terms: interventions — Fondaparinux

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Drug: Arixtra (fondaparinux), 2.5 mg/day-what is bioavailability

SUMMARY:
Patients in intensive care units have higher risks for developing blood clots. Arixtra inhibits blood clot formation by binding with the blood clotting factor, Xa. Critical illnesses and, specifically, medications given in the ICU to increase arterial blood pressure (vasopressors) may impair the absorption of drugs like Arixtra that are given subcutaneously. The study will measure the levels of Arixtra in blood comparing those subjects who are and those subjects who are not on blood pressure medication.

DETAILED DESCRIPTION:
In view of the high risk of venous thrombolism (VTE) in critically ill patients, it is essential for all ICUs to develop a standardized approach to thromboprophylaxis. Several studies in a critical setting have shown that both low dose unfractionated heparin and low molecular weight heparin (LMWH) reduce the incidence of VTE and either one of them is recommended as a valid agent by the newer ACCP consensus guidelines.

However, even with prophylaxis, critically ill patients still develop VTE. Common conditions amongst ICU patients such as generalized edema, poor peripheral perfusion during shock states, moderate renal dysfunction, etc., are possible explanations for this observation. Additionally, the use of vasoactive drugs may also impair peripheral circulation and reduce effective levels of agents used for the prevention of VTE.

This prospective clinical trial will be conducted to assess whether impaired peripheral circulation due to vasopressor (blood pressure) infusion decreases the bioavailability (i.e., plasma concentration) of subcutaneously administered fondaparinux (i.e., does vasopressor infusion lower blood plasma concentrations of fondaparinux), thereby reducing the prophylactic benefits of fondaparinux administration.

Fondaparinux (Arixtra®) was chosen as the anti-thrombotic agent to be used in this study because of its unique pharmacological properties and its safety and efficacy amongst different medical populations. Fondaparinux sodium administered by subcutaneous injection is rapidly and completely absorbed (absolute bioavailability is 100%). Following a single subcutaneous dose of fondaparinux sodium 2.5 mg in young male subjects, Cmax of 0.34 mg free acid/L is reached in approximately 2 hours. In patients undergoing treatment with fondaparinux sodium injection 2.5 mg, once daily, the peak steady-state plasma concentration is, on average, 0.39-0.50 mg free acid/L and is reached approximately 3 hours post-dose. Because fondaparinux does not react with platelet factor IV, thrombocytopenia is not an unwanted side effect.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients 18 or over, weight 50 kg or more in the ICU will be enrollment eligible. Pregnant women and those with neuraxial anesthesia, renal or liver problems, or BMI over 40 are not eligible.

Exclusion Criteria:

* Patients under 18, weight less than 50 kg, pregnant women and those with neuraxial anesthesia, renal or liver problems, or BMI over 40 are not eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-02; Study Completion 2010-01

CONTACTS AND LOCATIONS:
Overall Officials: M. Safwan Badr, MD, Study Chair — Wayne State University, Division of Pulmonary, Asthma, Critical Care, and Sleep Medicine
Locations (1):
- Harper University Hospital, ICU, Detroit, Michigan, United States